CLINICAL TRIAL: NCT02713789
Title: A Double-blind, Placebo-controlled, Parallel Design, Randomized, Phase 2A Clinical Trial Evaluating the Potential Activity and Safety of hMaxi-K Gene Transfer in Males With Erectile Dysfunction
Brief Title: Phase 2A Clinical Trial Evaluating the Potential Activity and Safety of hMaxi-K Gene for ED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Urovant Sciences GmbH (Industry)
Collaborators: Dasman Diabetes Institute (Other); Ion Channel Innovations (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ION04-ED
Record Dates: First submitted 2016-03-01; First posted 2016-03-21 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-07

CONDITIONS: Erectile Dysfunction
Keywords: ED
MeSH Terms: conditions — Erectile Dysfunction | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- hMaxi-K (Active Comparator): Single Treatment/ two escalating dose levels (8000 µg and 16,000 µg injection). In each dose level, 11 participants will receive hMaxi-K and 6 will receive placebo (only one injection per each participant)
  Interventions: Drug: hMaxi-K Single Treatment/ 2 escalating dose levels (8000 µg and 16000 µg injection)
- Placebo (PBS-20% sucrose) (Placebo Comparator): PBS-20% sucrose administered during two single treatment dose levels (8000 µg and 16000 µg) by injection (only one injection per each participant)
  Interventions: Drug: Placebo (PBS-20% sucrose)

INTERVENTIONS:
Drug: hMaxi-K Single Treatment/ 2 escalating dose levels (8000 µg and 16000 µg injection)
  Other Names: hMaxi-K; URO-902
  Arms: hMaxi-K
Drug: Placebo (PBS-20% sucrose)
  Other Names: Placebo
  Arms: Placebo (PBS-20% sucrose)

SUMMARY:
To evaluate the safety and efficacy of a single intracavernous injection of hMaxi K (8000 µg and 16000 µg) or placebo upon penile rigidity or erection in males with erectile dysfunction longer than six months that is attributable to an underlying, stable medical condition.

DETAILED DESCRIPTION:
This study is a double-blind, placebo controlled, parallel design, Phase 2A study evaluating the potential activity and safety of a single administration of hMaxi-K (8000 or 16000 µg) or placebo (PBS sucrose 20%) injected into the corpus cavernosum of the penis in men who have been unable to tolerate, do not wish to continue, or have had unsuccessful results with, prior therapy for ED.

The study population is men with erectile dysfunction attributable to an underlying, stable medical condition but who are otherwise in good health. The target population is men with erectile dysfunction and those who have been unable to tolerate, do not wish to continue, or have had unsuccessful results with, prior therapy for ED and with an erectile function domain score of IIEF < 21 at screening and baseline.

Following screening and study drug administration at Week 0 (Visit 2 [V2]), eligible participants will be evaluated at Weeks 1 (V3), 4 (V4), 8 (V5), 12 (V6), and 24 (V7). At each study visit, participants will have a physical examination including examination of the penis (all visits), vital signs, electrocardiogram (ECG) (all visits). Laboratory evaluations including chemistry and hematology will be done at V1, V3, V4, V6, and V7. Urinalysis will be done V1, V2 (prior to dosing), V3, V4, V6, and V7. Endocrine parameters and PTT, PT, sed rate and CRP will be evaluated at V1, V3, and V7. The participant will complete the erectile function domain of the IIEF and Sexual Encounter Profile (SEP) at screening/baseline and at V2, (SEP and IIEF at V2 prior to dosing) V3, V4, V5, V6, and V7. In all participants, plasma specimens will be collected to assay for the presence of hSlo DNA by PCR (V2-V7). These will be kept frozen at -20°C or less at the site for eventual assay by Sponsor.

The primary efficacy outcome measures will include the Erectile Function (EF) domain of the International Index of Erectile Function (IIEF), Sexual Encounter Profile (SEP), Questions 2 and 3 from SEP. The IIEF EF domain has a 30-point total score, where higher scores reflect better erectile function. SEP is a diary in which participants record each sexual attempt made throughout the study. The two questions from the Sexual Encounter Profile (SEP) deal with the ability to achieve vaginal penetration (SEP2), and the ability to maintain an erection long enough for successful intercourse (SEP3). The erectile function domain category of the IIEF will be used to evaluate the change in erectile status from baseline following administration of hMaxi-K. Change from baseline on the six questions of the IIEF's Erectile function domain category at every visit after administration of study drug will be calculated and compared among the two dose and one placebo groups.

Safety will be assessed by analysis of adverse experiences, and abnormal findings on clinical laboratory tests, electrocardiogram, and physical examinations.

6 months per participant (approximately 2 years to enroll all participants)

A total of 35 participants were planned to be enrolled; N=11 on 8000 µg; N=11 on 16000 µg; N=13 on placebo.

Both the safety data and data to assess activity will be presented as means and standard deviations or medians and ranges as appropriate for continuous data, and analyzed using either paired t- or Wilcox on Sign Rank tests for within group changes, and with mixed effects or marginal models to determine differences in trends among the three cohorts over time. Incidence of adverse events will be presented as relative frequencies within groups.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants must meet the following inclusion criteria:

  1. Signed Informed Consent
  2. Be adult males over 18 years of age diagnosed with erectile dysfunction and whose ED is attributable to an underlying, stable medical condition such as hypertension and atherosclerosis, antihypertensive medication, type I and type II diabetes mellitus, pelvic surgery and pelvic radiation, cerebrovascular accidents (stroke), multiple sclerosis, and Parkinson's disease;
  3. Participants must have been unable to have successful sexual intercourse for 3 months prior to study entry without specific ED therapy such as Vacuum Erection device (VED), ViagraTM (sildenafil), Cialis TM (tadalafil), MuseTM (alprostadil), or intracavernous injection therapy with an erectile function domain score of IIEF<21 at screening and baseline;
  4. Have been unable to tolerate, do not wish to continue, or have had unsuccessful results with, prior therapy for ED, e.g., ViagraTM, intracavernous injection therapy, MuseTM, or VED;
  5. If diabetic, documentation of HgA1c less than or equal to 8.0% prior to enrollment;
  6. If receiving medication for hypertension, documentation of blood pressure has been stable on the same medication for at least 2 months prior to enrollment;
  7. Be heterosexual and in a stable, monogamous relationship of at least six months duration;
  8. Agree to attempt intercourse with their partner at least four times per month while participating in the study;
  9. Agree not to use other treatments for ED while participating in this study;
  10. Have screening laboratory values and ECG that are within the normal range. See exclusion criterion below.
  11. A prior penile prosthetic implant;
  12. Have a normal physical examination of the penis;
  13. If participant had a radical prostatectomy a PSA <0.4 for at least one year documented by 2 measurements during the preceding year;
  14. Be literate, able to give written informed consent, and comply with all study procedures and requirements.

Exclusion Criteria:

1. A history of sickle-cell disease, sickle cell trait, or any other medical condition that, in the judgment of the investigator, would contraindicate the administration of study medication or interfere with the study evaluations;
2. In the judgment of the investigator any condition that would interfere with participation in the study (including geographical inaccessibility), that would contraindicate the administration of study medication or interfere with the study evaluations.
3. Had within six months prior to enrollment any of the following:

   * Myocardial infarction
   * Cerebrovascular accident
   * Uncontrolled hypertension (systolic >160 or diastolic >100mmHg)
   * Arrhythmia
   * Congestive heart failure (dyspnea on minimal exertion or while supine)
   * Unstable angina (chest pain greater than three times weekly while on therapy)
   * Required treatment with calcium channel, beta-blocker medication, nitrates, or anti-epileptic drugs;
4. Poorly controlled diabetes mellitus as defined by HgA1c > 8.0 mg% at time of enrollment;
5. Change in medication for diabetes or hypertension within 2 months of study enrollment;
6. Gonadal failure (testosterone < 200 ng/dl) not treated with hormone replacement;
7. History of malignancy except non-melanomatous skin cancers;
8. A life expectancy of less than 12 months;
9. An indwelling urethral catheter;
10. A prior penile prosthetic implant;
11. Received an investigational drug, investigational therapy, or other form of ED therapy, including approved treatments, within the past 30 days;
12. Peyronie's disease;
13. Any screening laboratory values outside of the normal laboratory range as defined by the central laboratory normal ranges and in the judgment of the investigator is considered clinically significant (hepatic biochemical markers [AST, ALT, GGT, alkaline phosphatase, and bilirubin] > twice the upper limit of the normal reference range may be accepted with written consent of the sponsor).
14. Any clinically significant ECG abnormality

NOTE: Sinus bradycardia of 50-59 bpm is permissible. Other abnormalities that can be normal variants (and considered clinically insignificant) may be permissible. However, participants with such abnormalities cannot be randomized without review of their medical history and prior written approval of the sponsor (or designee).

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-04; Primary Completion 2017-08-24 (Actual); Study Completion 2017-08-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Dasman, Kuwait

IPD SHARING:
Plan to Share IPD: Yes
publication

RESULTS

PARTICIPANT FLOW:
Groups:
- hMaxi-K 8000 µg: Participants received a single injection of hMaxi-K 8000 micrograms (µg) into the corpus cavernosum of the penis.
- hMaxi-K 16000 µg: Participants received a single injection of hMaxi-K 16000 µg into the corpus cavernosum of the penis.
- Placebo: Participants received a single injection of matching placebo (PBS-20% sucrose) into the corpus cavernosum of the penis.
Period: Overall Study
Arm/Group | hMaxi-K 8000 µg | hMaxi-K 16000 µg | Placebo
Started | 8 | 10 | 8
Completed | 8 | 9 | 7
Not Completed | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | hMaxi-K 8000 µg | hMaxi-K 16000 µg | Placebo | Total
Number analyzed (Participants) | 8 | 10 | 8 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (7.32) | 59.7 (9.2) | 59.1 (6.31) | 58.3 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 8 | 10 | 8 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Middle Eastern | 7 | 10 | 8 | 25
  Asian | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Experiences as Measured by Changes in Physical Examination of the Penis
Description: Physical examination of the penis included inspection and palpation.
Time Frame: up to Week 24 ± 3 days
Population: Safety Population: all participants who were randomized to any of the treatment groups and who have received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | hMaxi-K 8000 µg | hMaxi-K 16000 µg | Placebo
Number analyzed (Participants) | 8 | 10 | 8
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Significant Changes in Clinical Laboratory Parameters as Measured on Interval Blood and Urine Tests
Description: Clinical significance was determined by the Investigator using central laboratory values.
Time Frame: up to Week 24 ± 3 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | hMaxi-K 8000 µg | hMaxi-K 16000 µg | Placebo
Number analyzed (Participants) | 8 | 10 | 8
Participants | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Significant Changes on the Cardiogram as Measured by Significant Prolongation of QT Intervals and Cardiac Rhythm
Description: Clinical significance was determined by the Investigator using central laboratory values.
Time Frame: up to Week 24 ± 3 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | hMaxi-K 8000 µg | hMaxi-K 16000 µg | Placebo
Number analyzed (Participants) | 8 | 10 | 8
Participants | 0 | 2 | 0

4. Secondary Outcome: Mean Change From Baseline in the Percentage of "Yes" Responses to Questions 2 and 3 of the Sexual Encounter Profile (SEP) at Week 24
Description: SEP is a diary in which participants record each sexual attempt made throughout the study and is composed of 5 questions assessing sexual function. Two questions from the SEP deal with the ability to achieve vaginal penetration (Question 2: Were you able to insert your penis into your partner's vagina?), and the ability to maintain an erection (Question 3: Did your erection last long enough for you to have successful intercourse?). The number of "yes" response to each question in the SEP was computed as (Sum of all "yes" responses to respective SEP question /Total number of responses to that SEP question)*100. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 24
Population: Modified Intent-to-Treat (mITT) Population: all participants in the Intent-to-Treat (ITT) Population (all participants who were randomized to either of the treatment groups and who received at least one dose of study treatment) who had at least one post-dose efficacy assessment
Measure: Mean (95% Confidence Interval); unit: percentage of responses
Arm/Group | hMaxi-K 8000 µg | hMaxi-K 16000 µg | Placebo
Number analyzed (Participants) | 8 | 10 | 8
percentage of responses
  SEP2 | -18.8 [-47.78 to 10.28] | -16.7 [-57.45 to 24.12] | -28.6 [-73.70 to 16.56]
  SEP3 | -3.1 [-10.51 to 4.26] | 0 [0 to 0] | 0 [-53.40 to 53.40]
Statistical Analysis 1: Comparison: hMaxi-K 8000 µg vs Placebo; SEP2; Test type: Superiority; p = 0.827, ANCOVA
Statistical Analysis 2: Comparison: hMaxi-K 16000 µg vs Placebo; SEP2; Test type: Superiority; p = 0.594, ANCOVA
Statistical Analysis 3: Comparison: hMaxi-K 8000 µg vs Placebo; SEP3; Test type: Superiority; p = 0.274, ANCOVA
Statistical Analysis 4: Comparison: hMaxi-K 16000 µg vs Placebo; SEP3; Test type: Superiority; p = 0.766, ANCOVA

5. Secondary Outcome: Change From Baseline in the Erectile Function (EF) Domain of the International Index of Erectile Function (IIEF) at Week 24
Description: The IIEF is a validated, self-administered questionnaire that is a valid measure of male erectile dysfunction. The test contains 15 questions in 5 domains: (1) Erectile duration/function (questions [Q] 01 to 05 and 15); (2) Orgasmic function (questions 09 and 10); (3) Sexual desire (questions 11 and 12); (4) Intercourse satisfaction (questions 06, 07, and 08); (5) Overall sexual satisfaction (questions 13 and 14). The EF domain has been validated to assess erectile changes only. The domain-specific scores were calculated as the sum of the scores of the questions in the respective domain; thus, the total score of the EF domain was the sum of the 6 questions. Score range: 0 to 5 (Q01 to Q05), 1 to 5 (Q15). Total score: 1 to 30. Higher scores reflect better erectile function. Change from Baseline was calculated as the post-Baseline score minus the Baseline score.
Time Frame: Baseline; Week 24
Population: mITT Population. Only those participants with data available were analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | hMaxi-K 8000 µg | hMaxi-K 16000 µg | Placebo
Number analyzed (Participants) | 8 | 9 | 7
score on a scale | -0.9 (2.86) | -2.1 (1.85) | -5.3 (2.08)
Statistical Analysis 1: Comparison: hMaxi-K 8000 µg; Test type: Superiority; p = 0.384, t-test, 1 sided; one-sided paired t-test at 5% significance level
Statistical Analysis 2: Comparison: hMaxi-K 16000 µg; Test type: Superiority; p = 0.144, t-test, 1 sided; one-sided paired t-test at 5% significance level
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority; p = 0.022, t-test, 1 sided; one-sided paired t-test at 5% significance level
Statistical Analysis 4: Comparison: hMaxi-K 16000 µg vs Placebo; Test type: Superiority; p = 0.137, t-test, 1 sided; p-value (one-sided) corresponds to the two sample t-test analysis
Statistical Analysis 5: Comparison: hMaxi-K 8000 µg vs Placebo; Test type: Superiority; p = 0.123, t-test, 1 sided; p-value (one-sided) corresponds to the two sample t-test analysis

6. Secondary Outcome: Change From Baseline in the Orgasmic Function Domain of the International Index of Erectile Function (IIEF) at Week 24
Description: The IIEF is a validated, self-administered questionnaire that is a valid measure of male erectile dysfunction. The test contains 15 questions in 5 domains: (1) Erectile duration/function (questions 01 to 05 and 15); (2) Orgasmic function (questions 09 and 10); (3) Sexual desire (questions 11 and 12); (4) Intercourse satisfaction (questions 06, 07, and 08); (5) Overall sexual satisfaction (questions 13 and 14). The domain-specific scores were calculated as the sum of the scores of the questions in the respective domain; thus, the total score of the Orgasmic Function domain was the sum of 2 questions. Score range: 0 to 5 (Q09 and Q10). Total score: 0 to 10. Higher scores reflect better erectile function. Change from Baseline was calculated as the post-Baseline score minus the Baseline score.
Time Frame: Baseline; Week 24
Population: mITT Population. Only those participants with data available were analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | hMaxi-K 8000 µg | hMaxi-K 16000 µg | Placebo
Number analyzed (Participants) | 8 | 9 | 7
score on a scale | -1.5 (1.40) | 1.1 (1.30) | -0.3 (0.57)
Statistical Analysis 1: Comparison: hMaxi-K 8000 µg; Test type: Superiority; p = 0.160, t-test, 1 sided; one-sided paired t-test at 5% significance level
Statistical Analysis 2: Comparison: hMaxi-K 16000 µg; Test type: Superiority; p = 0.208, t-test, 1 sided; one-sided paired t-test at 5% significance level
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority; p = 0.316, t-test, 1 sided; one-sided paired t-test at 5% significance level
Statistical Analysis 4: Comparison: hMaxi-K 8000 µg vs Placebo; Test type: Superiority; p = 0.221, t-test, 1 sided; p-value (one-sided) corresponds to the two sample t-test analysis
Statistical Analysis 5: Comparison: hMaxi-K 16000 µg vs Placebo; Test type: Superiority; p = 0.172, t-test, 1 sided; p-value (one-sided) corresponds to the two sample t-test analysis

7. Secondary Outcome: Change From Baseline in the Sexual Desire Domain of the International Index of Erectile Function (IIEF) at Week 24
Description: The IIEF is a validated, self-administered questionnaire that is a valid measure of male erectile dysfunction. The test contains 15 questions in 5 domains: (1) Erectile duration/function (questions 01 to 05 and 15); (2) Orgasmic function (questions 09 and 10); (3) Sexual desire (questions 11 and 12); (4) Intercourse satisfaction (questions 06, 07, and 08); (5) Overall sexual satisfaction (questions 13 and 14). The domain-specific scores were calculated as the sum of the scores of the questions in the respective domain; thus, the total score of the Sexual Desire domain was the sum of 2 questions. Score range: 1 to 5 (Q11 and Q12). Total score: 2 to 10. Higher scores reflect better erectile function. Change from Baseline was calculated as the post-Baseline score minus the Baseline score.
Time Frame: Baseline; Week 24
Population: mITT Population. Only those participants with data available were analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | hMaxi-K 8000 µg | hMaxi-K 16000 µg | Placebo
Number analyzed (Participants) | 8 | 9 | 7
score on a scale | -0.9 (0.97) | -1.0 (1.14) | 0.0 (1.29)
Statistical Analysis 1: Comparison: hMaxi-K 8000 µg; Test type: Superiority; p = 0.199, t-test, 1 sided; one-sided paired t-test at 5% significance level
Statistical Analysis 2: Comparison: hMaxi-K 16000 µg; Test type: Superiority; p = 0.203, t-test, 1 sided; one-sided paired t-test at 5% significance level
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority; p = 0.500, t-test, 1 sided; one-sided paired t-test at 5% significance level
Statistical Analysis 4: Comparison: hMaxi-K 8000 µg vs Placebo; Test type: Superiority; p = 0.296, t-test, 1 sided; p-value (one-sided) corresponds to the two sample t-test analysis
Statistical Analysis 5: Comparison: hMaxi-K 16000 µg vs Placebo; Test type: Superiority; p = 0.286, t-test, 1 sided; p-value (one-sided) corresponds to the two sample t-test analysis

8. Secondary Outcome: Change From Baseline in the Intercourse Satisfaction Domain of the International Index of Erectile Function (IIEF) at Week 24
Description: The IIEF is a validated, self-administered questionnaire that is a valid measure of male erectile dysfunction. The test contains 15 questions in 5 domains: (1) Erectile duration/function (questions 01 to 05 and 15); (2) Orgasmic function (questions 09 and 10); (3) Sexual desire (questions 11 and 12); (4) Intercourse satisfaction (questions 06, 07, and 08); (5) Overall sexual satisfaction (questions 13 and 14). The domain-specific scores were calculated as the sum of the scores of the questions in the respective domain; thus, the total score of the Intercourse Satisfaction domain was the sum of 3 questions. Score range: 0 to 5 (Q06 through Q8). Total score: 0 to 15. Higher scores reflect better erectile function. Change from Baseline was calculated as the post-Baseline score minus the Baseline score.
Time Frame: Baseline; Week 24
Population: mITT Population. Only those participants with data available were analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | hMaxi-K 8000 µg | hMaxi-K 16000 µg | Placebo
Number analyzed (Participants) | 8 | 9 | 7
score on a scale | -0.1 (0.93) | -0.3 (1.07) | -2.3 (0.75)
Statistical Analysis 1: Comparison: hMaxi-K 8000 µg; Test type: Superiority; p = 0.449, t-test, 1 sided; one-sided paired t-test at 5% significance level
Statistical Analysis 2: Comparison: hMaxi-K 16000 µg; Test type: Superiority; p = 0.381, t-test, 1 sided; one-sided paired t-test at 5% significance level
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority; p = 0.011, t-test, 1 sided; one-sided paired t-test at 5% significance level
Statistical Analysis 4: Comparison: hMaxi-K 8000 µg vs Placebo; Test type: Superiority; p = 0.05, t-test, 1 sided; p-value (one-sided) corresponds to the two sample t-test analysis
Statistical Analysis 5: Comparison: hMaxi-K 16000 µg vs Placebo; Test type: Superiority; p = 0.09, t-test, 1 sided; p-value (one-sided) corresponds to the two sample t-test analysis

9. Secondary Outcome: Change From Baseline in the Overall Sexual Satisfaction Domain of the International Index of Erectile Function (IIEF) at Week 24
Description: The IIEF is a validated, self-administered questionnaire that is a valid measure of male erectile dysfunction. The test contains 15 questions in 5 domains: (1) Erectile duration/function (questions 01 to 05 and 15); (2) Orgasmic function (questions 09 and 10); (3) Sexual desire (questions 11 and 12); (4) Intercourse satisfaction (questions 06, 07, and 08); (5) Overall sexual satisfaction (questions 13 and 14). The domain-specific scores were calculated as the sum of the scores of the questions in the respective domain; thus, the total score of the Overall Sexual Satisfaction domain was the sum of 2 questions. Score range: 1 to 5 (Q13 and Q14). Total score: 2 to 10. Higher scores reflect better erectile function. Change from Baseline was calculated as the post-Baseline score minus the Baseline score.
Time Frame: Baseline; Week 24
Population: mITT Population. Only those participants with data available were analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | hMaxi-K 8000 µg | hMaxi-K 16000 µg | Placebo
Number analyzed (Participants) | 8 | 9 | 7
score on a scale | -1.1 (0.69) | 0.1 (1.34) | -1.11 (0.83)
Statistical Analysis 1: Comparison: hMaxi-K 8000 µg; Test type: Superiority; p = 0.074, t-test, 1 sided; one-sided paired t-test at 5% significance level
Statistical Analysis 2: Comparison: hMaxi-K 16000 µg; Test type: Superiority; p = 0.468, t-test, 1 sided; one-sided paired t-test at 5% significance level
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority; p = 0.109, t-test, 1 sided; one-sided paired t-test at 5% significance level
Statistical Analysis 4: Comparison: hMaxi-K 8000 µg vs Placebo; Test type: Superiority; p = 0.493, t-test, 1 sided; p-value (one-sided) corresponds to the two sample t-test analysis
Statistical Analysis 5: Comparison: hMaxi-K 16000 µg vs Placebo; Test type: Superiority; p = 0.235, t-test, 1 sided; p-value (one-sided) corresponds to the two sample t-test analysis

10. Secondary Outcome: Mean Change From Baseline in the Percentage of "Yes" Responses to Questions 1, 4, and 5 of the Sexual Encounter Profile (SEP) at Week 24
Description: SEP is a diary in which participants record each sexual attempt made throughout the study and is composed of 5 questions assessing sexual function. Question 1: Were you able to achieve at least some erection?; Question 4: Were you satisfied with the hardness of your erection?; Question 5: Overall, were you satisfied with the sexual experience? The number of "yes" response to each question in the SEP was computed as (Sum of all "yes" responses to respective SEP question /Total number of responses to that SEP question)*100. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 24
Population: mITT Population
Measure: Mean (95% Confidence Interval); unit: percentage of responses
Arm/Group | hMaxi-K 8000 µg | hMaxi-K 16000 µg | Placebo
Number analyzed (Participants) | 8 | 10 | 8
percentage of responses
  SEP1 | 15.6 [-35.49 to 66.74] | -31.0 [-80.04 to 18.14] | -50.0 [-96.24 to -3.76]
  SEP4 | 12.5 [-17.06 to 42.06] | 14.3 [-20.67 to 49.24] | 0 [0 to 0]
  SEP5 | 0 [0 to 0] | 28.6 [-16.56 to 73.70] | 0 [0 to 0]
Statistical Analysis 1: Comparison: hMaxi-K 8000 µg vs Placebo; SEP1; Test type: Superiority; p = 0.136, ANCOVA
Statistical Analysis 2: Comparison: hMaxi-K 16000 µg vs Placebo; SEP1; Test type: Superiority; p = 0.498, ANCOVA
Statistical Analysis 3: Comparison: hMaxi-K 8000 µg vs Placebo; SEP4; Test type: Superiority; p = 0.369, ANCOVA
Statistical Analysis 4: Comparison: hMaxi-K 16000 µg vs Placebo; SEP4; Test type: Superiority; p = 0.337, ANCOVA
Statistical Analysis 5: Comparison: hMaxi-K 16000 µg vs Placebo; SEP5; Test type: Superiority; p = 0.160, ANCOVA

ADVERSE EVENTS:
Time Frame: Up to Week 24 (± 3 days)
Arm/Group | hMaxi-K 8000 µg | hMaxi-K 16000 µg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/10 | 1/8
Other Adverse Events (participants affected / at risk) | 8/8 | 10/10 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | hMaxi-K 8000 µg (N=8) | hMaxi-K 16000 µg (N=10) | Placebo (N=8)
Eye operation (Eye disorders) | 1 | 0 | 0
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | hMaxi-K 8000 µg (N=8) | hMaxi-K 16000 µg (N=10) | Placebo (N=8)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 0
Blood testosterone decreased (Investigations) | 0 | 2 | 1
Electrocardiogram QT prolonged (Investigations) | 2 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 8 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 3 | 4 | 0
Haematuria (Renal and urinary disorders) | 1 | 3 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT02713789/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT02713789/SAP_001.pdf